CLINICAL TRIAL: NCT02363244
Title: A Pilot Study on Comparative Evaluation of Results of Pap Smears and HPV Hybrid Capture 2 Performed on Cervical Samples Before and After Application of Acetic Acid
Brief Title: Pap and HPVDNA Before and After Acetic Acid
Status: Completed | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Gauravi Ashish Mishra, Associate Professor Dept of Preventive Oncology, Tata Memorial Hospital
Other Study IDs: 1413 Pap HPV Project
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: CIN
Keywords: Pap,HPVDNA

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — HPV DNA TEST will be collected in stored as per protocol of storage and will be analysed by hybridisation method in microbiologt Dept of Tata Memorial hospital.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pap group: Per speculum examination will be done.Pap test will be collected for the women as per allotement.A via (visual inspection with acedic acid)test will be done.A repeat cervical cell for pap test will be collected and send to laboratory for further evaluation.
- HPVDNA GROUP: Per speculum examination will be done.HPVDNA test will be collected for the women as per allotement.A via (visual inspection with acedic acid)test will be done.A repeat cervical cell for HPVDNA will be collected and send to laboratory for further evaluation.

SUMMARY:
This is a pilot study to assess the cell adequacy and quality of Pap smears and adequacy of samples for HPV DNA virus test done after application of 5%acetic acid in a VIA test.Normally a Pap test and HPV DNA test is performed before application of acetic acid. It is assumed that application of acetic acid may alter the cell adequacy of Pap test and HPV DNA test, if any of the above tests is done immediately after VIA test.The present study aims to see the effect of 4-5% acetic acid [vinegar] on the cell adequacy and quality of Pap smear and sample adequacy for HPV DNA test.

DETAILED DESCRIPTION:
Aim (of pilot study):

To evaluate the cell adequacy and smear quality of Pap smears and adequacy of samples for HPV HC 2 collected before and after application of acetic acid.

Objective of Pilot study-

1. Agreement between the results of HC2 on cervical samples obtained from women before and 5 to 10 mins after VIA test
2. Correlation between RLU/ cutoff ratio of HC2 on cervical samples obtained from women before and 5 to 10 mins after VIA test.
3. Agreement between the results of cytology on cervical smears obtained immediately before and 5 to 10 mins after VIA test from the same women.

Methodology:

Design: Pilot study

Study Duration: Three months

Study Site: Preventive Oncology screening clinic, Tata Memorial Hospital

Sample Size calculation and power estimates:

For the pilot study, sampling method is a convenience sample of 50 consecutive eligible women attending the Preventive Oncology screening clinic and consenting to participate in the study. These women will be randomly allocated using lottery method (wherein 25 chits with HPV and 25 chits with cytology written inside will be placed). For every participant woman a chit will be picked up and the woman will be allotted to either HPV or cytology testing depending on the message in the chit. Thereafter the chit will be discarded.

In 25 samples Pap smears will be collected before and after application of acetic acid. Steps mentioned below.

In rest 25 samples HPV DNA will be collected before and after application of acetic acid. Steps mentioned below.

Step 1: A per speculum examination will be performed on eligible women attending the Preventive Oncology screening clinic and the findings of the same will be recorded.

Step 2: Pap smear will be collected - Smear 1. OR Cervical cell samples will be collected for HPV HC II - HPV sample 1. Step 3: VIA will be performed and the findings will be noted. Step 4: A second Pap smear will be collected 5 to 10 minutes after performing VIA when the woman is still on the examination table by the same provider- Smear 2.

OR Cervical cell samples will be collected for HPV HC II - HPV sample 2. Step 5: The smears will be submitted to the cytology department for evaluation. The HPV HC II samples will be submitted to the Microbiology department for evaluation.

Step 6: The cytologist reading the smear will be blinded as to which smear was taken before and which was taken after the application of acetic acid. The same cytologist will read the pre-VIA and the post-VIA smears.

Similarly, the Microbiology department staff will be blinded as to which HPV sample was taken before and which was taken after the application of acetic acid. The paired samples will be analyzed at the same laboratory in the same batch of testing.

Step 7: The screen negative women will undergo routine follow-up. The screen positive women will undergo Colposcopy, guided biopsy and further management according to the Tata Memorial Hospital protocol.

Analysis of the variables Data entry will be done in the Department of Preventive Oncology, Tata Memorial Hospital using SPSS version 18. Checks for consistency, data safety and analysis will be carried out at regular intervals. Both descriptive and inferential statistics will be generated for describing variables under the study objectives. Agreement in HC2 results between pre-VIA and post-VIA samples will be estimated using kappa statistics. Similarly, agreement in pap results between pre-VIA and post-VIA samples will be estimated using kappa statistics. Sensitivity and specificity of HC2 test and pap test in detecting CIN2+ lesions will be calculated using negative colposcopy or biopsy as the gold standard and will be compared between the pre and post VIA samples.

ELIGIBILITY:
Inclusion Criteria:

* Married women attending the Preventive Oncology screening clinic.
* women in age group 30 to 60 years

Exclusion Criteria

* Unmarried women
* married women in the age group less than 30 years and above 60 years
* pregnant women
* women with history of total hysterectomy
* women with cervical cancer

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Married women attending the Preventive Oncology screening clinic in the age group 30 to 60 years for cervical cancer screening.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Comparative Evaluation Of Results Of Pap Smears And HPV Hybrid Capture 2 Performed On Cervical Samples Before And After Application Of Acetic Acid. | 3 months
  The purpose of this pilot study is to assess the cell adequacy and quality of Pap smears and adequacy of samples for HPV DNA virus test done after application of acetic acid.

CONTACTS AND LOCATIONS:
Overall Officials: Gauravi A Mishra,, MD, Principal Investigator — Tata Memorial Centre

REFERENCES:
- See also: Tata Memorial Centre, Mumbai Official website — http://tmc.gov.in